CLINICAL TRIAL: NCT01778595
Title: Pilot Study of the Fecal Microbiome in the Shanghai Population
Brief Title: Colon Cancer Study of Fecal Samples in Shanghai, China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Shanghai Center for Disease Control and Prevention (Other); BGI, China (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913068; 13-C-N068
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-09-21

CONDITIONS: Colorectal Neoplasms
Keywords: Microbiome; Feces; Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Early detection of colon cancer can improve the chances of successful treatment for most people. This approach is especially important if blood is detected in the stool. However, much better stool sample tests are needed to find this cancer early. To improve the tests, researchers want to collect samples from people who are already being screened for colon cancer. This study will collect information and samples from older adults in Shanghai, China. These adults will be participating in screening tests for colon cancer.

Objectives:

- To collect samples and medical information for colon cancer screening from older adults in Shanghai, China.

Eligibility:

* Adults between 50 and 74 years of age who are being screened for colon cancer.
* Participants will be recruited from two community health centers in Shanghai, China.

Design:

* Participants will provide information on their medical history and factors related to colon cancer. They will respond to questions on use of medications, diet choices (such as eating red meat), bowel habits, and other factors.
* Participants will collect samples for study. These samples will be collected within 3 days of the screening visit. Particpants will provide a urine sample and four stool samples. They will also use cotton swabs to collect samples from just inside the anus. The samples will be returned to the study doctors for research tests that may indicate who has colon cancer.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
To examine how risk for colorectal cancer (CRC) is related to the microbes that inhabit the distal human intestine (the microbiota), we have proposed a large study that compares characteristics of the fecal microbiota in CRC patients and controls in the Shanghai population. In advance of that, we are proposing a small pilot study with the following two objectives: 1) determine participation rates among Shanghai adults, age 50-74 who are positive by fecal immunochemical test (FIT+); and 2) determine the suitability of fecal specimens provided by the participants for microbiome analyses. Each of two Shanghai community health centers, where CRC screening is ongoing, will recruit 25 FIT+ participants (half male; half age 50-64, half age 65-74). Each of the 50 participants will provide informed consent, brief questionnaire data, blood plasma and buffy coat, a urine specimen, and four samples of one stool, which will be frozen. Complete blood count and plasma glucose, cholesterol, and creatinine levels will be determined in real time and returned to the participant. Each participant s plasma, buffy coat, urine, and one pair of fecal samples will be stored frozen for future genetic or other assays. DNA will be extracted from the second pair of fecal samples from each participant (n=100 vials), amplified for 16S rRNA genes, and sequenced to determine fecal microbiome profiles. Participation will be deemed unsatisfactory if participation is <30% overall (95% confidence interval 17% - 43% for N=50 participants), or if there are <20 male, female, younger, or older participants. Specimen quality will be deemed unsatisfactory if the intraclass correlation coefficient (ICC) is <0.70 (95% confidence interval 0.53 0.82 for N=50 paired vials) for the Shannon index estimate of microbiome alpha diversity. As amended, the two community health centers will recruit up to 600 additional adults presenting for CRC screening, irrespective of FITstatus, who will be asked to provide saliva as well as the other specimens.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Participation is restricted to adults age 50-74 who are: 1) residents of the catchment areas of the community health centers in Shanghai s Minhang and Xuhui Districts, and 2) are participating in the CRC screening program at those centers. Patients who do not provide signed informed consent will be excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-01-08; Primary Completion 2015-12-09 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Participation rate, data quality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James J Goedert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Shanghai Center for Disease Control and Prevention, Shanghai, China

REFERENCES:
- [Background] Arthur JC, Perez-Chanona E, Muhlbauer M, Tomkovich S, Uronis JM, Fan TJ, Campbell BJ, Abujamel T, Dogan B, Rogers AB, Rhodes JM, Stintzi A, Simpson KW, Hansen JJ, Keku TO, Fodor AA, Jobin C. Intestinal inflammation targets cancer-inducing activity of the microbiota. Science. 2012 Oct 5;338(6103):120-3. doi: 10.1126/science.1224820. Epub 2012 Aug 16. PMID 22903521
- [Background] Caporaso JG, Lauber CL, Walters WA, Berg-Lyons D, Huntley J, Fierer N, Owens SM, Betley J, Fraser L, Bauer M, Gormley N, Gilbert JA, Smith G, Knight R. Ultra-high-throughput microbial community analysis on the Illumina HiSeq and MiSeq platforms. ISME J. 2012 Aug;6(8):1621-4. doi: 10.1038/ismej.2012.8. Epub 2012 Mar 8. PMID 22402401
- [Background] Goedert JJ, Gong Y, Hua X, Zhong H, He Y, Peng P, Yu G, Wang W, Ravel J, Shi J, Zheng Y. Fecal Microbiota Characteristics of Patients with Colorectal Adenoma Detected by Screening: A Population-based Study. EBioMedicine. 2015 Apr 18;2(6):597-603. doi: 10.1016/j.ebiom.2015.04.010. eCollection 2015 Jun. PMID 26288821